CLINICAL TRIAL: NCT03876210
Title: A Randomized, Open-label, Single Dose, 2x2 Crossover Phase 1 Clinical Trial to Evaluate the Safety and Pharmacokinetic Characteristics After Administration of Fixed-dose Combination or Loose Combination of PK101 in Healthy Volunteers
Brief Title: Study to Compare the Safety and Pharmacokinetics of PK101 With Coadministration of the Two Separate Drugs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PMG Pharm Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PK101_P102
Record Dates: First submitted 2019-03-13; First posted 2019-03-15 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Other): Period 1: PK101-001, PK101-002 / Period 2: PK101
  Number of subject: 23
  Wash out Period: over 7 days (between each period)
  Dosage: Once daily, at 2D each period
  Interventions: Combination Product: PK101; Drug: PK101-001, PK101-002
- Sequence B (Other): Period 1: PK101 / Period 2: PK101-001, P101-002
  Number of subject: 23
  Wash out Period: over 7 days (between each period)
  Dosage: Once daily, at 2D each period
  Interventions: Combination Product: PK101; Drug: PK101-001, PK101-002

INTERVENTIONS:
Combination Product: PK101 — PK101-001 + PK101-002 (combination)
Drug: PK101-001, PK101-002 — coadministration

SUMMARY:
The purpose of this study is to compare the safety and pharmacokinetics of PK101(fixed-dose combination of PK101-001 and PK101-002) with coadministration of the two separate drugs in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults ≥ 19 years of age (on the day of screening)
* Body weigth ≥50.0kg, 18.5Kg/(m)^2 ≤ (BMI) ≤30.0Kg/(m)^2
* No congenital or chronic diseases and no abnormal signs determined by medical examinations
* Not abnormal or not clinical significant lab values
* Understand the requirements of the study and voluntarily consent to participate in the study.

Exclusion Criteria:

* Clinically significant disease with liver, renal, neurologic, respiratory, digestive, endocrine, hemato-oncology, urologic, cardiovascular, musculoskeletal, psychiatric system
* Subjects who have hypersensitivity for investigational products
* AST or ALT > 2*ULN, r-GTP > 1.5*ULN, Blood creatinine > ULN (ULN, Upper Limit of Normal)
* SBP ≥ 140 mmHg or< 90 mmHg, DBP ≥ 90 mmHg or < 60 mmHg
* Subjects who were administered below medications within 30 days (barbiturates, drugs of induced or suppressive drug metabolizing enzyme, etc)
* Subjects who previously participated in other clinical trials or bioequivalence Test within 6 months
* Subjects with whole blood donation within 2 months or component blood donation within 1 month or blood transfusion within 1 month prior to the first dosing.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
AUCt | 0(Pre-dose), 0.5, 1, 1.5, 2, 2.33, 2.67, 3, 3.5, 4, 6, 8, 12, 24, 36, 48 hour
  Area under the plasma/serum/blood drug concentration-time curve from time zero to the time of the last quantifiable concentration of PK101-002
Cmax | 0(Pre-dose), 0.5, 1, 1.5, 2, 2.33, 2.67, 3, 3.5, 4, 6, 8, 12, 24, 36, 48 hour
  Maximum Plasma Concentration of PK101-002

SECONDARY OUTCOMES:
Tmax | 0(Pre-dose), 0.5, 1, 1.5, 2, 2.33, 2.67, 3, 3.5, 4, 6, 8, 12, 24, 36, 48 hour
  Time of peak concentration of PK101-002
AUCinf | 0(Pre-dose), 0.5, 1, 1.5, 2, 2.33, 2.67, 3, 3.5, 4, 6, 8, 12, 24, 36, 48 hour
  Area under the plasma concentration versus time curve from zero to infinity of PK101-002
t1/2 | 0(Pre-dose), 0.5, 1, 1.5, 2, 2.33, 2.67, 3, 3.5, 4, 6, 8, 12, 24, 36, 48 hour
  Terminal half life of PK101-002
CL/F | 0(Pre-dose), 0.5, 1, 1.5, 2, 2.33, 2.67, 3, 3.5, 4, 6, 8, 12, 24, 36, 48 hour
  Clearance/Bioavailability of PK101-002
AUCt/AUCinf | 0(Pre-dose), 0.5, 1, 1.5, 2, 2.33, 2.67, 3, 3.5, 4, 6, 8, 12, 24, 36, 48 hour
  AUCt/AUCinf of PK101-002

CONTACTS AND LOCATIONS:
Overall Officials: Jang-Hee Hong, Principal Investigator — Clinical Trials Center, Chungnam National University Hospital
Locations (1):
- Clinical Trials Center, Chungnam National University Hospital, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Song JH, Koh H, Moon HY, Jung JG, Hong JH, Sunwoo J. Comparison of a fixed-dose combination of Celecoxib/PG201 [Layla(R)] versus co-administration of individual formulations in healthy participants: A randomized trial. Medicine (Baltimore). 2024 Nov 15;103(46):e40494. doi: 10.1097/MD.0000000000040494. PMID 39560548